CLINICAL TRIAL: NCT01692093
Title: KM110329 in Adult Patients With Atopic Dermatitis : a Randomised, Double-blind, Placebo-controlled, Multicenter Trial
Brief Title: KM110329 in Adult Patients With Atopic Dermatitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kyunghee University Medical Center (Other)
Collaborators: St Mary's Hospital, London (Other); Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other); Kyung Hee University Hospital at Gangdong (Other)
Responsible Party: Principal Investigator, Seong-Gyu Ko, Professor, Kyunghee University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CCRG_KM110329
Record Dates: First submitted 2012-09-17; First posted 2012-09-25 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-11

CONDITIONS: Atopic Dermatitis
Keywords: SCORAD; Atopic dermatits; Skin health
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- KM110329 (Experimental): Participants will receive KM110329 for eight weeks. Participants will take 2 tablets by mouth with water two times a day after meals.
  Interventions: Dietary Supplement: KM110329
- Control (Placebo Comparator): Participants will receive placebo drug for eight weeks. Participants will take 2 tablets by mouth with water two times a day after meals.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: KM110329 — KM110329, a functional food consist of four herbs which are shown to be beneficial for skin health
  Arms: KM110329
Dietary Supplement: Placebo — Placebo
  Arms: Control

SUMMARY:
The purpose of this study is to determine clinical efficacy and safety of KM110329 for Atopic dermatitis.

DETAILED DESCRIPTION:
A randomized, double blind, placebo-controlled, multicenter trial will be conducted at the Seoul St.Mary's Hospital, at Chung-ang University hospital, and at Kyung Hee University Hospital at Gangdong.

Participants fulfilling eligibility criteria will be selected. Enrolled participants will be randomly allocated to two parallel groups: the KM110329 and placebo arms.

Each participant will be examined for signs and symptoms of Atopic dermatitis before and after taking functional food.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 18 to 65 years
* Individuals who diagnosed Atopic dermatitis according to the criteria of Hanifin and Rajka
* Individuals who mild to moderate atopic dermatitis (objective SCORAD≤40)
* Written informed consent for participation in the trial

Exclusion Criteria:

* Severe skin disease other than Atopic dermatitis
* Secondary infection with bacteria, fungi, and virus
* Uncontrolled hypertension (SBP > 145 mmHg or DBP > 95 mmHg)
* Severe liver disability (2.5-fold the normal high range value for ALT, AST)
* Severe renal disability (sCr > 2.0mg/dl)
* Women who are pregnant, lactating, planning a pregnancy or women of child-bearing age who do not agree to proper contraception
* Use of oral steroids, oral antibiotic or other immunosuppressants within the past 4 weeks
* Treated by systemic photochemotherapy within past 4 weeks
* History of drug abuse
* Hypersensitivity to Rubi Fructus, Houttuyniae Herba, Rehmanniae Radix, Betulae Platyphyllae Cortex
* Use of other investigational products within the past two months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2012-09; Primary Completion 2014-06 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
SCORAD index | 8 weeks
  SCORing Atopic Dermatitis

SECONDARY OUTCOMES:
DLQI | 8 weeks
  The Dermatology Life Quality Index

OTHER OUTCOMES:
TEWL | 8 weeks
  Transepidermal Water Loss
hydration in the stratum corneum | 8 weeks
  hydration in the stratum corneum
KiFDA-HM-AD | 8 weeks
  Evaluation endpoint for clinical trial of herbal medicinal products about atopic dermatitis

CONTACTS AND LOCATIONS:
Overall Officials: SEONG GYU KO, M.D.(DKM), Study Director — Kyunghee University
Locations (1):
- Kyung Hee University, Seoul, South Korea

REFERENCES:
- [Derived] Cheon C, Park S, Park JS, Oh SM, Jang S, Go HY, Jang BH, Shin YC, Ko SG. KM110329 in adult patients with atopic dermatitis: a randomised, double-blind, placebo-controlled, multicentre trial--study protocol. BMC Complement Altern Med. 2013 Nov 27;13:335. doi: 10.1186/1472-6882-13-335. PMID 24279519